CLINICAL TRIAL: NCT03472209
Title: Comparison of Different EtCO2 Levels in Preventing Postoperative Nausea and Vomiting in Gynecological Patients Undergoing Laparoscopic Surgery
Brief Title: Comparison of Different EtCO2 Levels in Preventing Postoperative Nausea and Vomiting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ahmet Besir, Assistant professor, Karadeniz Technical University
Other Study IDs: 2017/237
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Gynecological Laparoscopic Surgery; End-tidal carbon dioxide
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: ETCO2=26-35 mmHg
- Group B: ETCO2=36-45 mmHg

SUMMARY:
We aimed to evaluate the different ETCO2 levels (with the help of ultrasonographic optic nerve sheath diameter) in preventing gynecological laparoscopic surgeons' postoperative nausea induced by intracranial pressure change due to pneumoperitoneum and trandelenburg position.

DETAILED DESCRIPTION:
Although gynecologic laparoscopic surgery is a preferred technique in recent years due to its minimally invasive technique, the incidence of postoperative nausea and vomiting (PONV) is 53-72%. In such operations, intra-abdominal pressure due to trandelenburg position and carbondioxide insufflation causes intra-cranial venous obstruction and intra-cranial pressure increase. In addition, intra-cranial blood flow and ultimately intra-cranial pressure increase due to gravity and increased venous return resistance (peripheral vascular resistance). Intra-cranial CO2 concentration increase results in intra-cranial vascular dilatation, followed by ICP increase. High intracranial pressure may cause an increase in the incidence of PONV after gynecological laparoscopic surgery. Measurement of optic nerve sheath diameter with USG, a noninvasive method for detecting intracranial pressure increases, has been used frequently in intensive care units in recent years. we aimed to evaluate the different ETCO2 levels (during the operation with 10 minute intervals, and also with the help of ultrasonographic optic nerve sheath diameter) in preventing gynecological laparoscopic surgeons' postoperative nausea induced by intracranial pressure change due to pneumoperitoneum and trandelenburg position.

ELIGIBILITY:
Inclusion Criteria:

25-50 age, ASA I / II, BMI: 18-33 kg/m2, operation time: 50-130 min., gynecological laparoscopy

Exclusion Criteria:

In previous operations, Patients with postoperative nausea-vomiting (PONV) history, Smoking, Vehicle stays, Liver and kidney dysfunction, Abnormal fluid electrolyte balance, Gastrointestinal system disease, Preoperative antiemetic drug use, Cerebral disease,dysrhythmia

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with gynecological laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
EtCO2 | During the operation (in 10 minutes interval)
  End tidal carbondioxide

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Besir, MD, Study Chair — Karadeniz Teknit Üniversitesi Tıp Fakültesi
Locations (2):
- Turkey (Türkiye) (2):
  - Karadeniz Teknik Universitesi, Trabzon
  - Karadeniz Technical University, Dept Obs and Gyn / Anestesiology, Trabzon